## **Statistical Plan**

Official Title: Visceral Manipulation in Patients With Chronic Low Back Pain

NCT03101020

**Document Date**: November, 18th 2016

## **Statistical Analysis Plan**

Intention to treat analysis was employed when necessary, with the data from the previous evaluation repeated to substitute missing data. The Kolmogorov-Sirmonov test demonstrated normal data distribution. Thus, parametric tests were performed and the data were expressed as mean and standard deviation. Two-way analysis of variance (ANOVA) was used to compare the effects of stimulation during motor training on the main outcome variables and the Bonferroni correction for multiple comparisons was employed as the post hoc test. The dependent variables were pain intensity, lumbar mobility, general functionality and specific functionality. The independent fixed variables were treatment (baseline, posttreatment and follow-up), group (experimental group and control group) and group—treatment interaction. The Pearson correlation test verified the correlation between the outcomes of the variables. A p-value <0.05 indicated a statistically significant result. The data were organized and tabulated using the Statistical Package for Social Sciences (v.19.0).